CLINICAL TRIAL: NCT02528786
Title: A Phase 1, Single-Time Blood Sample Collection Study for Pharmacogenomic Characterization of Subjects That Previously Received Namilumab and Participated in the Phase 1 PRIORA Study
Brief Title: Blood Sample Collection Study for Pharmacogenomic Characterization of Participants That Previously Received Namilumab in M1-1188-002-EM (PRIORA, [NCT01317797]) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Namilumab-1003; 2015-000571-27 (EudraCT Number); U1111-1168-0946 (Registry Identifier: UTN (WHO)); NL53485.058.15 (Registry Identifier: CCMO)
Record Dates: First submitted 2015-08-13; First posted 2015-08-19 (Estimated); Results first posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Drug therapy
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- All Participants (Other): Participants who received namilumab previously in M1-1188-002-EM (PRIORA, [NCT01317797]) will have blood samples collected on Day 1.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No study drug will be administered in this study.

SUMMARY:
The purpose of this study is to obtain blood samples from up to 14 participants who previously received namilumab in the previous study M1-1188-002-EM (PRIORA, [NCT01317797]) to correlate genetic markers with clinical outcomes.

DETAILED DESCRIPTION:
Participants who received treatment with namilumab in the previous study M1-1188-002-EM (PRIORA [NCT01317797]) will have two whole blood samples (3 mL each) collected to correlate genetic markers with namilumab treatment responses as determined in the previous study.

The study will enroll approximately 14 participants who received namilumab in the previous study.

• No intervention is administered in this study.

This trial will be conducted in Bulgaria, Spain and The Netherlands. The overall time to participate in this study is 1 day.

ELIGIBILITY:
Inclusion Criteria:

1. The participant (or, when applicable, the participant's legally acceptable representative) voluntarily signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

1. Did not receive namilumab during the PRIORA study (A phase Ib double-blind, placebo controlled, randomized, dose-escalating study).
2. Participants without any response time point recorded 4-week after the last dose of namilumab and beyond this time point
3. Participants who were excluded from post-hoc analysis due to protocol violations during the previous PRIORA study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2016-04-05 (Actual); Study Completion 2016-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in The Netherlands, Bulgaria, and Spain from 19 November 2015 to 05 April 2016.
Pre-assignment Details: Participants with a historical diagnosis of mild or moderate rheumatoid arthritis who received namilumab (MT203) in the study M1-1188-002-EM (NCT01317797) were enrolled in this study to obtain and analyze a blood deoxyribonucleic acid (DNA) sample.
Groups:
- All Participants: Participants who received namilumab in the phase 1 PRIORA M1-1188-002-EM (NCT01317797) were enrolled. Two blood samples (3 milliliter [mL] per sample) for DNA isolation were collected from each participant.
Period: Overall Study
Arm/Group | All Participants
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The analysis set included all participants who were enrolled and completed the study.
Groups:
- All Participants: Participants who received namilumab in the phase 1 PRIORA M1-1188-002-EM (NCT01317797) were enrolled. Two blood samples (3 mL per sample) for DNA isolation were collected from each participant.
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Customized [Number; unit: participants]
  Adults (18-64 years) | 5
  Adults (65-84 years) | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race/Ethnicity, Customized [Number; unit: participants]
  White | 8
Region of Enrollment [Number; unit: participants]
  Netherlands | 3
  Bulgaria | 4
  Spain | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Each Cluster
Description: Clusters are described by an ellipse whose major and minor axes are the standard deviations in the x and y directions of the component points, which are rotated so that their covariance is equal to zero. The clusters were based upon the algorithms in which each data-point is assigned to one of four clusters: 1, 2, 3, or 4, representing no-target (negative controls [NTCs]), homozygotes one (XX), homozygotes two (YY), and heterozygotes (XY), respectively. Based on the calculated genetic composite scores from 8-single-nucleotide polymorphism (SNP)-based algorithm, participants were segregated into clusters.
Time Frame: Baseline
Population: The analysis set included all participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 8
participants
  Cluster 1 | 0
  Cluster 2 | 4
  Cluster 3 | 4
  Cluster 4 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 166
Description: No deaths, serious adverse events (SAE) or other significant adverse events (AE) were reported. The risk in this study was only related to blood draws since no drug was ever administered.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.